CLINICAL TRIAL: NCT03702101
Title: Detecting Auricular Points Among Patients With Orofacial Pain by A Novel Auricular Point Detector (APD): A Pilot Diagnostic Accuracy Study
Brief Title: Detecting Auricular Points in OFP by a Novel APD ( APD-OFP)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); City University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: SCM-ACU-02
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Orofacial Pain
Keywords: orofacial pain; auricular point; electrical impedance
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orofacial pain group: Patients in this group will receive auricular point detection which is accomplished by the novel auricular point detector device. There is no addition to the patient's routine care.
  Interventions: Device: Auricular point detector
- Control group: This group includes healthy subject, for whom no treatment will be performed. Only auricular point detection by the auricular point detector will be conducted.
  Interventions: Device: Auricular point detector

INTERVENTIONS:
Device: Auricular point detector — This device is only for auricular detection. No additional intervention will be delivered.

SUMMARY:
This is a pilot diagnostic accuracy study conducted to assess the diagnostic ability of a novel APD for auricular point detection among patients with orofacial pain, as compared with an already commercialized device.

DETAILED DESCRIPTION:
The present study is a pilot diagnostic accuracy study conducted to assess the diagnostic ability of a novel APD for auricular point detection among patients with orofacial pain (OFP), as compared with an already commercialized device. This study will examine if the novel APD is more reliable than the traditional devices currently available in the market. Moreover, this study will also use the APD device to test the cutaneous electrical impedance of the ear and further assess whether the orofacial auricular points is with the lowest electrical impedance in the OFP population. This pilot study will enroll 12 OFP patients from the Department of Anesthesiology, Queen Mary Hospital, the University of Hong Kong. 12 healthy subjects will be recruited as control from the university community. Auricular acupoint detection will be accomplished with the new device and a control device. The electrical impedance will be detected and recorded. Patient's condition will also be evaluated by the Penn Facial Pain Scale-Revised (2018). The specificity and sensitivity of the auricular point detection by the APD device will be calculated. Cohen's kappa coefficient (κ) will be used to test the inter-methods reliability, test-retest reliability, and inter-tester reliability. Moreover, the Pearson Correlation Coefficient will be used to test the correlation between the electrical impedance of the auricular point of the orofacial area and the Penn Facial Pain Scale score.

ELIGIBILITY:
Inclusion Criteria:

* When pain attacks, the average unilateral orofacial pain severity >=5 point measured by a 10-point VAS scale;
* Patient with trigeminal neuralgia can be diagnosed according to Trigeminal neuralgia: New classification and diagnostic grading for practice and research (Neurology, 2016);
* Other kinds of orofacial pain can be diagnosed based on the patient's symptoms;
* Provide written inform consent;
* Free of any other diagnosed psychological conditions;

Exclusion Criteria:

* with any other diseases such as cardiovascular, renal, neurological, digestive, hepatic, respiratory disease;
* Pregnancy or lactation;
* Participation in a clinical study that may interfere with participation in this study;
* History of or current tobacco, alcohol use;
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study;
* Unable to provide written informed consent due to any reason;

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: OFP patients visiting the inpatient or outpatient unit of the Department of Anesthesiology Queen Mary Hospital will be referred to this study by an anesthesiologist.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
cohen's kappa coefficient | baseline
  The Cohen's kappa coefficient is a statistical test used to validate the inter-method reliability, test-retest reliability and inter-observer reliability of the device in detecting OFP-related auricular point.

SECONDARY OUTCOMES:
the Visual Analogue Scale (VAS) | baseline
  The VAS is a common instrument used to measure pain intensity. The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates worst pain possible.
the Penn Facial Pain Scale-Revised (Penn-FPS-R) | baseline
  The Penn-FPS-R is a new 12-item Health-Related Quality of Life outcome measure with content validity that can be used to assess and monitor the impact of Trigeminal Neuralgia and facial pain treatment interventions in both clinical practice and research. This scale uses the 0-10 numeric rating scale (NRS) to quantify the pain intensity and its impact on life quality, where 0 indicates no pain/impact and 10 indicates worst pain/impact. The sum of the rated NRS score will be calculated.
self-developed questionnaire on patient's attitude towards complementary therapies for pain management | baseline
  This is a self-developed questionnaire which includes 10 items aiming to survey patient's attitude towards the use of complementary therapies for pain management. This questionnaire only includes descriptive answers to be choose. The percentage for each choice will calculated.
The diagnostic specificity of the device | baseline
  The specificity test is a test to validate the ability of a diagnosis to tell the 'non-disease' among those without the disease.
The diagnostic sensitivity of the device | baseline
  The sensitivity test is a test to validate the ability of a diagnosis to tell the 'disease' among those with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lixing Lao, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, HKU, Hong Kong, INTL, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be at the discretion of the study-involved participants and the principal investigator.